CLINICAL TRIAL: NCT07161713
Title: Pilot Study of a Social/Behavioral Intervention on Lung, Colon, and Non-Hodgkin's Lymphoma (NHL) Cancer Survivors, Evaluating the Effect of Mind Body Interventions on Patient Reported Outcomes, Inflammation and Epigenetics.
Brief Title: SBU-RESET: RElaxation, Stress Reduction and Epigenetics Trial in Cancer Survivors
Acronym: RESET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Nemesure (Other)
Responsible Party: Sponsor-Investigator, Barbara Nemesure, Professor, Department of Family, Population and Preventive Medicine, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-RESET; IRB2025-00282 (Other: Stony Brook University)
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Lung Adenocarcinoma; Lung Adenocarcinoma Metastatic; Lung Adenocarcinoma Stage III; Lung Adenocarcinoma Stage IIIB/IV; Lung Adenocarcinoma Stage IV; Lung Adenocarcinoma Stage I; Lung Adenocarcinoma Stage II; NHL; NHL - Non-Hodgkin&Amp;#39;s Lymphoma; Lung Cancer (Diagnosis); Colon Cancer
Keywords: stony brook; survivor; yoga; mindfulness-based stress reduction; holistic
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms; Disease; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial pilot study, with a within-subject lead-in control period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): Oncology-informed yoga
  Interventions: Behavioral: Oncology-informed yoga
- SMART (Experimental): Stress Management and Resiliency Training
  Interventions: Behavioral: SMART

INTERVENTIONS:
Behavioral: Oncology-informed yoga — 8 weekly sessions of cancer informed-yoga incorporating light movement, breathing techniques, and some meditation practices
  Arms: Yoga
Behavioral: SMART — SMART, developed by the Impact Foundation, is an adaptation of Mindfulness-based Stress Reduction (MBSR) approach that incorporates other elements like mindful self-compassion, emotional literacy, and positive psychology principles to address the unique stressors faced by teachers.
  Arms: SMART

SUMMARY:
Cancer survivors can experience health issues that cause chronic illness and lower quality of life. Yoga is a well-known holistic approach to health and overall well-being. Mindfulness has many benefits, including improved focus and less stress. This study aims to evaluate if yoga and/or mindfulness has a positive effect on cancer survivors social, emotional and physical well-being as well as their epigenetics. Epigenetics is how the environment can effect your genes; not by changing our DNA, but by turning genes on or off.

DETAILED DESCRIPTION:
Randomized interventional pilot study to evaluate whether a mind-body intervention (Stress Management and Resiliency Training (SMART) or (oncology-informed yoga) influences patient-reported Quality of life (QoL) outcomes (physical/social/emotional/ functional well-being and symptom burden) in Lung Colon, and Non-Hodgkin's lymphoma (NHL) survivors. A secondary (exploratory) aim is to evaluate whether these mind-body interventions impact epigenetics.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Primary diagnosis: Lung Cancer, Colon Cancer and Non-Hodgkin's lymphoma (NHL)
* Six months post cancer-directed treatment (chemotherapy, targeted and immunotherapy). Patients with active disease (e.g. metastatic colorectal cancer) who are not receiving any cancer-directed treatment are eligible.
* Able to provide a saliva sample
* Gives informed consent and agrees to be randomly assigned
* Able to complete the questionnaire(s) in English.

Exclusion Criteria:

* Adults with primary anal and/or primary rectal cancer.
* Adult cancer survivors who are currently on an active treatment regimen.
* Oral or any pathological conditions that can limit the ability to produce saliva.
* Unable to participate in full length study period and follow up thereafter.
* Is pregnant or plan to become pregnant during the study period.
* Currently practicing yoga or SMART
* Those on corticosteroid therapy.
* Documented fall or syncope within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2027-09-17 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Quality of Life by EORTC QLQ-C30 | 8 weeks
  Patient reported quality of life measured using the quality of life questionnaire C30 (QLQ-C30), developed by the European Organisation for Research and Treatment of Cancer. This scale includes 5 functional and 3 symptom scales, each scored as a 0-100 scale, where higher scores indicate a better outcome on functional scales and global health status, and a worse outcome on symptoms.
Patient Reported Quality of Life by QLQ-CR29 | 8 weeks
  Patient (colon cancer only) reported quality of life measured using the quality of life questionnaire (QLQ-CR29), developed by the European Organisation for Research and Treatment of Cancer. This scale is a validated 29-item symptom scale used in conjunction with the core EORTC QLQ-C30 questionnaire, to assess the quality of life of patients with colon and rectal cancer. Note: rectal cancer is an exclusion criteria. An estimate of the average of the items in the scale is the raw score. The raw score is linearly transformed to a 0-100-point range with higher scores indicating a higher ("better") level of functioning or a higher ("worse") level of symptoms. An estimate of the average of the items in the scale is the raw score. The raw score is linearly transformed to a 0-100-point range with higher scores indicating a higher ("better") level of functioning or a higher ("worse") level of symptoms
Patient Reported Quality of Life by QLQ-LC29 | 8 weeks
  Patient (lung cancer only) reported quality of life measured using questionnaire QLQ-LC29, developed by the European Organisation for Research and Treatment of Cancer. This is a validated, 29-item questionnaire used in conjunction with the core EORTC QLQ-C30 questionnaire to assess the quality of life of patients with lung cancer. An estimate of the average of the items in the scale is the raw score. The raw score is linearly transformed to a 0-100-point range with higher scores indicating a higher ("better") level of functioning or a higher ("worse") level of symptoms
Patient Reported Quality of Life by QLQ-NHL-HG29 | 8 weeks
  Patient (high-grade non-Hodgkins lymphoma cancer only) reported quality of life measured using questionnaire QLQ-NHL-HG29, a 29-item health-related quality of life questionnaire developed by the European Organisation for Research and Treatment of Cancer (EORTC) for patients with high-grade non-Hodgkin lymphoma (HG-NHL). It is used in conjunction with the core EORTC QLQ-C30 questionnaire to assess health-related quality of life, including aspects of symptom burden, physical condition, fatigue, emotional impact, and worries about health, which allows for better evaluation of treatments. An estimate of the average of the items in the scale is the raw score. The raw score is linearly transformed to a 0-100-point range with higher scores indicating a higher ("better") level of functioning or a higher ("worse") level of symptoms
Patient Reported Quality of Life by QLQ-NHL-LG20 | 8 weeks
  Patient (low-grade non-Hodgkins lymphoma cancer only) reported quality of life measured using questionnaire QLQ-NHL-LG29, a 20-item health-related quality of life questionnaire developed by the European Organisation for Research and Treatment of Cancer (EORTC) for patients with low-grade non-Hodgkin lymphoma (LG-NHL). It is used in conjunction with the core EORTC QLQ-C30 questionnaire to assess health-related quality of life, including aspects of symptom burden, physical condition, fatigue, emotional impact, and worries about health, which allows for better evaluation of treatments. An estimate of the average of the items in the scale is the raw score. The raw score is linearly transformed to a 0-100-point range with higher scores indicating a higher ("better") level of functioning or a higher ("worse") level of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Nemesure, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Cancer Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No